CLINICAL TRIAL: NCT05180877
Title: Asthma During Pregnancy; Impact of Asthma Severity
Brief Title: Asthma During Pregnancy; Impact of Severity
Status: Completed | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Hend Mohammed Abdelraheem Esmaeel, assistant professor, Sohag University
Other Study IDs: Soh-Med-21-09-35
Record Dates: First submitted 2021-11-20; First posted 2022-01-06 (Actual); Last update posted 2022-01-06 (Actual); Status verified 2021-12

CONDITIONS: Bronchial Asthma
Keywords: Bronchial asthma; Asthma; pregnancy; Asthma severity
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intermittent& mild persistent asthma: According to asthma severity assessment, this group included asthmatic pregnant females patients with intermittent asthma and mild persistent asthma
- Moderate& severe persistent asthma: According to asthma severity assessment, this group included asthmatic pregnant females patients with Moderate& severe persistent asthma

SUMMARY:
bronchial asthma (BA) may affect pregnancy and this affection may increase with increasing asthma severity. This study was designed to detect the effect of asthma severity on the course of asthma during pregnancy and its effect on the pregnancy and perinatal outcome

DETAILED DESCRIPTION:
This was prospective study conducted in sohag university hospital ( obstetric outpatient clinic, chest outpatient clinic and emergency department ).This study aimed to detect the effect of baseline asthma severity on the course of asthma during pregnancy and its effect on the pregnancy and perinatal outcome in the setting of advancements in the management and pharmacotherapy of asthma compared with that previously

ELIGIBILITY:
Inclusion Criteria:

* pregnant women in ages 18y or more with confirmed diagnosis of bronchial asthma presenting in1st trimester to inpatient or outpatients clinic of chest department.

Exclusion Criteria:

* Patients with Chest diseases other than bronchial asthma and patients with cardiac disease.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — pregnant asthmatic women
Study Population: Pregnant asthmatic female patients presenting in first trimester to inpatient or outpatients clinic of chest department.
Sampling Method: Probability Sample
Enrollment: 137 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
maternal complications | from the start of inclusion to the study till termination of pregnancy, average 9 months period
  Occurrence any pregnancy related complication to the parturient women was recorded in both study groups.
perinatal complications | from the start of inclusion to the study till termination of pregnancy, average 9 months period
  Incidence of any fetal or neonatal complication was recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dharmage SC, Perret JL, Custovic A. Epidemiology of Asthma in Children and Adults. Front Pediatr. 2019 Jun 18;7:246. doi: 10.3389/fped.2019.00246. eCollection 2019. PMID 31275909
- [Background] Robijn AL, Murphy VE, Gibson PG. Recent developments in asthma in pregnancy. Curr Opin Pulm Med. 2019 Jan;25(1):11-17. doi: 10.1097/MCP.0000000000000538. PMID 30407268
- [Background] National Asthma Education and Prevention Program. Expert Panel Report 3 (EPR-3): Guidelines for the Diagnosis and Management of Asthma-Summary Report 2007. J Allergy Clin Immunol. 2007 Nov;120(5 Suppl):S94-138. doi: 10.1016/j.jaci.2007.09.043. PMID 17983880